CLINICAL TRIAL: NCT01285830
Title: Primary Prevention of Allergic Disease in Early Child by Lactobacillus Reuteri
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Collaborators: BioGaia AB (Industry); The Ekhaga Foundation, Sweden (Unknown); The Heart and Lung foundation, Sweden (Unknown); The Research Council for the South-East Sweden (Unknown); The Swedish Asthma and Allergy Association, Sweden (Unknown); The Swedish Research Council (Other Government); University Hospital, Linkoeping (Other)
Responsible Party: Professor Bengt Björkstén, The National Institute of Environmental Medicine, Karolinska Institutet, Stockholm, Sweden
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BGB 99/02; F2000-106 (Other Grant/Funding Number: Research Council for the South-East Sweden)
Record Dates: First submitted 2011-01-27; First posted 2011-01-28 (Estimated); Last update posted 2014-03-20 (Estimated); Status verified 2011-01

CONDITIONS: Allergic Conditions
Keywords: Infants; Probiotics; Prevention; Lactobacillus reuteri; Eczema; IgE; Sensitization; Microbiota; Chemokines
MeSH Terms: conditions — Eczema

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo
- Lactobacillus reuteri (Active Comparator)
  Interventions: Dietary Supplement: Lactobacillus reuteri

INTERVENTIONS:
Dietary Supplement: Lactobacillus reuteri — The mothers started taking Lactobacillus reuteri ATCC 55730 (BioGaia AB, Stockholm, Sweden) or placebo four weeks before term and continued to do so daily until delivery. After birth, the baby commenced with the same study product as the mother at 1-3 days of age and continued daily for one year. The daily intake, five oil droplets, corresponded to 1 x 100 000 000 colony forming units (CFU)
  Arms: Lactobacillus reuteri
Dietary Supplement: Placebo — The placebo consists of the same oil that the active study product but without any bacteria and is not possible to differentiate from the active product by smell, taste or visual appearance
  Arms: Placebo

SUMMARY:
An altered microbial exposure may be partly responsible for the increase of allergic diseases in populations with a western lifestyle. Activation of the immune system by microbes early in life is probably required for an accurate maturation of the immune system. Probiotics, live bacteria which are considered to confer health when ingested, have been suggested to prevent eczema and sensitisation infants.

The aim of this study is to assess the effect of oral supplementation with the probiotic bacterium Lactobacillus reuteri in infancy on the development of allergic disease and sensitisation during the first 2 years of life and to examine mechanisms possibly underlying eventual effects on allergic manifestations.

A follow up was performed at 7 years of age.

DETAILED DESCRIPTION:
An altered microbial exposure may be partly responsible for the increase of allergic diseases in populations with a western lifestyle. Activation of the immune system by microbes early in life is probably required for an accurate maturation of the immune system. Probiotics, live bacteria which are considered to confer health when ingested, have been suggested to prevent eczema and sensitisation infants.

The aim of this study is to assess the effect of oral supplementation with the probiotic bacterium Lactobacillus reuteri (L. reuteri) in infancy on the development of allergic disease and sensitisation during the first 2 years of life and to examine mechanisms possibly underlying eventual effects on allergic manifestations. In the study the development of allergic disease will also be related prospectively to immunological, nutritional and environmental factors.

The study is a prospective double-blind placebo-controlled multicenter trial, comprising 232 families with allergic disease. The families are recruited at the antenatal clinic, and the mothers will receive L. reuteri ATCC 55730 (1 x 100 000 000 colony forming units, Biogaia AB, Stockholm, Sweden) or placebo daily from gestational week 36 until delivery. Their babies then will continue with the same study product from birth until 12 months of age and will be followed up for another year. Clinical follow-up will be done at 1, 3, 6,12 and 24 months of age and telephone interviews at 2,4,5, 8, 10 and 18 months. A questionnaire will be completed on each occasion. Skin prick test will be performed at 6, 12 and 24 months of age. Venous blood will be collected from the umbilical cord and at 6, 12 and 24 months and stored as heparinized plasma or serum until assessment. Peripheral mononuclear blood cells (PBMC) will be separated from the plasma samples before storage. Blood samples will also be collected from the mother and father once during the study. The stool sample will be collected from the mother during the 1 week after delivery and the infant at 5-7 days, 1 month, 3 months, 6 months, 12 months and 24 months of age. Saliva samples will be collected at 3, 6, 12 and 24 months of age and breast milk samples will be collected from the mother 1-3 days and 1 months after delivery. The saliva, breast milk and plasma/serum samples will be stored in -20°C and stool samples and the PBMC in -70°C until assessment.

A follow up was performed at 7 years of age focusing on allergic disease. Spirometry, skin prick test was performed. Of the 188 completing the 2 year follow up, 184 also completed the 7 year follow up.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with history of previous or present allergic disease in at least one member of the immediate family (parents or siblings).
* Expected compliance.
* Written informed consent obtained from parents.

Exclusion Criteria:

* Insufficient compliance, i.e. a consumption of the study product below half of the expected.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2001-02; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Allergic disease | Incidence until 2 years of age
  Allergic disease was defined as any of the following: eczema, asthma, allergic rhinoconjunctivitis, allergic urticaria, gastrointestinal allergy. These diagnosis are based on predefined criteria.

SECONDARY OUTCOMES:
Sensitization | incidence until 2 years of age
  Positive skin prick test and /or circulation IgE against allergen in blood
IgE-associated allergic disease | Incidence until 2 years of age
  Allergic disease was classified as IgE-associated if the symptomatic infant also was sensitized
Lactobacillus reuteri colonization in stool and breast milk | Point prevalance until 2 years of age
  Isolation of Lactobacillus reuteri in stool and breast milk samples from the mother and infant with conventional and molecular methods.
Cytokines in breast milk | 1-3 days and 1 months postpartum
  Cytokines in breast milk from the mother will be measured by ELISA.
Th1 and Th2- associated chemokines in blood samples | Development from birth until 2 years of age
  Th1 and Th2- associated chemokines will be analyzed in blood samples from the infant with ELISA and Luminex.
Microbial composition in stool samples | Development from birth until 2 years of age
  The microbial composition in stoll samples from the mothers and infants will be assessed with conventional cultivation and molecular microbiology methods
Allergic disease at 7 years of age | 2001-2011
  Allergic disease at 7 years of age was defined as any of the following: eczema, asthma, allergic rhinoconjunctivitis, allergic urticaria. These diagnosis are based on predefined criteria.
Prevalence of caries in primary dentition at 8 years of age | 2009-2012
  Prevalence of caries in primary dentition is examined by dentists at 8 yeas of age. These diagnosis are based on predefined criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Bengt Björkstén, MD, PhD, Principal Investigator — The National Institute of Environmental Medicine, Karolinska Institutet, Stockholm, Sweden
Locations (3):
- Sweden (3):
  - Pediatric Clinic, Ryhov Hospital, Jönköping
  - Pediatric Clinic, University Hospital, Linköping
  - Pediatric Clinic, Vrinnevi Hospital, Norrköping

REFERENCES:
- [Result] Abrahamsson TR, Jakobsson T, Bottcher MF, Fredrikson M, Jenmalm MC, Bjorksten B, Oldaeus G. Probiotics in prevention of IgE-associated eczema: a double-blind, randomized, placebo-controlled trial. J Allergy Clin Immunol. 2007 May;119(5):1174-80. doi: 10.1016/j.jaci.2007.01.007. Epub 2007 Mar 8. PMID 17349686
- [Result] Bottcher MF, Abrahamsson TR, Fredriksson M, Jakobsson T, Bjorksten B. Low breast milk TGF-beta2 is induced by Lactobacillus reuteri supplementation and associates with reduced risk of sensitization during infancy. Pediatr Allergy Immunol. 2008 Sep;19(6):497-504. doi: 10.1111/j.1399-3038.2007.00687.x. Epub 2008 Jan 22. PMID 18221472
- [Result] Abrahamsson TR, Sinkiewicz G, Jakobsson T, Fredrikson M, Bjorksten B. Probiotic lactobacilli in breast milk and infant stool in relation to oral intake during the first year of life. J Pediatr Gastroenterol Nutr. 2009 Sep;49(3):349-54. doi: 10.1097/MPG.0b013e31818f091b. PMID 19525871
- [Result] Connolly E, Abrahamsson T, Bjorksten B. Safety of D(-)-lactic acid producing bacteria in the human infant. J Pediatr Gastroenterol Nutr. 2005 Oct;41(4):489-92. doi: 10.1097/01.mpg.0000176179.81638.45. No abstract available. PMID 16205524
- [Result] Abrahamsson TR, Sandberg Abelius M, Forsberg A, Bjorksten B, Jenmalm MC. A Th1/Th2-associated chemokine imbalance during infancy in children developing eczema, wheeze and sensitization. Clin Exp Allergy. 2011 Dec;41(12):1729-39. doi: 10.1111/j.1365-2222.2011.03827.x. Epub 2011 Aug 1. PMID 21801246
- [Result] Abrahamsson TR, Jakobsson HE, Andersson AF, Bjorksten B, Engstrand L, Jenmalm MC. Low diversity of the gut microbiota in infants with atopic eczema. J Allergy Clin Immunol. 2012 Feb;129(2):434-40, 440.e1-2. doi: 10.1016/j.jaci.2011.10.025. Epub 2011 Dec 6. PMID 22153774
- [Result] Forsberg A, Abrahamsson TR, Bjorksten B, Jenmalm MC. Pre- and post-natal Lactobacillus reuteri supplementation decreases allergen responsiveness in infancy. Clin Exp Allergy. 2013 Apr;43(4):434-42. doi: 10.1111/cea.12082. PMID 23517039
- [Result] Jakobsson HE, Abrahamsson TR, Jenmalm MC, Harris K, Quince C, Jernberg C, Bjorksten B, Engstrand L, Andersson AF. Decreased gut microbiota diversity, delayed Bacteroidetes colonisation and reduced Th1 responses in infants delivered by caesarean section. Gut. 2014 Apr;63(4):559-66. doi: 10.1136/gutjnl-2012-303249. Epub 2013 Aug 7. PMID 23926244
- [Result] Abrahamsson TR, Jakobsson T, Bjorksten B, Oldaeus G, Jenmalm MC. No effect of probiotics on respiratory allergies: a seven-year follow-up of a randomized controlled trial in infancy. Pediatr Allergy Immunol. 2013 Sep;24(6):556-61. doi: 10.1111/pai.12104. Epub 2013 Jul 31. PMID 23902407
- [Result] Abrahamsson TR, Jakobsson HE, Andersson AF, Bjorksten B, Engstrand L, Jenmalm MC. Low gut microbiota diversity in early infancy precedes asthma at school age. Clin Exp Allergy. 2014 Jun;44(6):842-50. doi: 10.1111/cea.12253. PMID 24330256
- [Derived] Forsberg A, Abrahamsson TR, Bjorksten B, Jenmalm MC. Pre- and postnatal administration of Lactobacillus reuteri decreases TLR2 responses in infants. Clin Transl Allergy. 2014 Jun 25;4:21. doi: 10.1186/2045-7022-4-21. eCollection 2014. PMID 25002964
- [Derived] Abrahamsson TR, Rautava S, Moore AM, Neu J, Sherman PM. The time for a confirmative necrotizing enterocolitis probiotics prevention trial in the extremely low birth weight infant in North America is now! J Pediatr. 2014 Aug;165(2):389-94. doi: 10.1016/j.jpeds.2014.05.012. Epub 2014 Jun 16. No abstract available. PMID 24948349